CLINICAL TRIAL: NCT07309718
Title: MRI-Derived Pressure Ratio: a Novel Noninvasive Hemodynamic Biomarker for Stroke Risk Stratification in Intracranial Atherosclerotic Stenosis
Brief Title: MPR for Stroke Risk Assessment of ICAS
Status: Recruiting | Type: Observational
Sponsor: Xuanwu Hospital, Beijing (Other)
Collaborators: Xuanwu Hebei Hospital (Unknown); Xuanwu Xiongan Hospital (Unknown); Xuanwu Chifeng Hospital (Unknown); Xuanwu Jinan Hospital (Unknown)
Responsible Party: Sponsor
Other Study IDs: CASSISS-MPR
Record Dates: First submitted 2025-12-15; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: ICAS - Intracranial Atherosclerosis; Stroke Ischemic; Hemodynamic
Keywords: ICAS - Intracranial Atherosclerosis; Stroke Ischemic; Hemodynamic; Pressure ratio
MeSH Terms: conditions — Intracranial Arteriosclerosis; Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CASSISS-MPR
  Interventions: Drug: Standardized medical therapy targeting vascular risk factors and stroke prevention

INTERVENTIONS:
Drug: Standardized medical therapy targeting vascular risk factors and stroke prevention — Dual antiplatelet treatment and management of vascular risk factors, in accordance with AHA/ASA guidelines

SUMMARY:
Intracranial atherosclerotic stenosis (ICAS) carries substantial stroke risk despite optimal medical treatment. Current risk stratification relies primarily on stenosis severity, but novel hemodynamic markers may improve prediction. In this multiple prospective registry study we aim to investigate whether regional hemodynamics, measured by a novel Magnetic resonance imaging-derived Pressure Ratio (MPR) technique, are associated with stroke risk in ICAS.

DETAILED DESCRIPTION:
This study is a multicentre prospective single-arm registry study and the protocol is approved by the ethics committee at the coordinating centre and by the local institutional review board at each participating centre. This study is initiated by the investigators, with 5 participating stroke centres , and plans to recruit 400 consecutive patients who meet the inclusion and exclusion criteria. After the enrolment, all participants would be evaluated at baseline, 1 month, 6 months, and 12 months post-enrollment. All participants received standardized medical therapy, including dual antiplatelet treatment and management of vascular risk factors, in accordance with AHA/ASA guidelines. Multimodal imaging techniques were employed to assess hemodynamic status: luminal stenosis would be evaluated using transcranial Doppler (TCD), computed tomography angiography (CTA), magnetic resonance angiography (MRA), or digital subtraction angiography (DSA), high-resolution MRI and phase-contrast MR angiography (PC-MRA) would be collected to calculate MPR. The primary outcomes were ischemic stroke in the qualifying artery territory or related death within 1 year. There were 5 secondary outcomes, including hemodynamic ischemic stroke in the qualifying artery territory within1 year. An independent Data and Safety Monitoring Board (DSMB) oversees the conduction, safety and efficacy of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18 to 80 years.
2. Intracranial atherosclerotic stenosis ICAS involving a culprit artery in the anterior circulation.
3. Intracranial arterial stenosis of 50% to 99% as measured by the WASID method using TCD, CTA, MRA, or DSA.
4. Written informed consent obtained from the participant or a legal representative.

Exclusion Criteria:

1. Non-atherosclerotic intracranial lesions, including moyamoya disease, vasculitis, vascular dissection, autoimmune diseases, or congenital/genetic abnormalities.
2. More than 50% stenosis of the extracranial carotid artery on the ipsilateral side.
3. Large cerebral infarction involving more than one-half of the territory on DWI imaging, or a baseline modified Rankin Scale score ≥3.
4. Contraindications to antiplatelet therapy or statins.
5. Inability to undergo MRI due to metal implants or claustrophobia.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with ICAS involving 50% to 99% stenosis of a major intracranial artery in the anterior circulation, including the internal carotid artery (ICA C6-C7 segment) and the middle cerebral artery M1 (MCA-M1) segment.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2027-12-15 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
ischemic stroke in the qualifying artery territory or related death within 1 year after enrollment. | 12 months
  the number of participants who suffer from ischemic stroke in the qualifying artery territory or related death within 1 year after enrollment.

SECONDARY OUTCOMES:
transient ischemic attack (TIA) or ischemic stroke in the qualifying artery territory within 1 year | 12 months
  the number of participants who suffer from transient ischemic attack (TIA) or ischemic stroke in the qualifying artery territory within 1 year after enrollment.
TIA related to ischemia in the qualifying artery territory within 1 year | 12 months
  the number of participants who suffer from TIA related to ischemia in the qualifying artery territory within 1 year
any stroke/TIA/ death within 1 year | 12 months
  the number of participants who suffer from any stroke/TIA/ death within 1 year
hemodynamic ischemic stroke in the qualifying artery territory within 1 year | 12 months
  the number of participants who suffer from hemodynamic ischemic stroke in the qualifying artery territory within 1 year
embolic stroke within in the qualifying artery territory 1 year | 12 months
  the number of participants who suffer from embolic stroke within in the qualifying artery territory 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurosurgery, Xuanwu hospital, Beijing, Xicheng District, China

IPD SHARING:
Plan to Share IPD: No